CLINICAL TRIAL: NCT04796909
Title: A Parent-Coaching Intervention to Promote Community Participation of Young Children With Developmental Disability
Brief Title: Occupational Performance Coaching With Parents of Young Children With Developmental Disability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Food and Health Bureau, Hong Kong (Other Government); University of Otago (Other); National Cheng Kung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZC2Q
Record Dates: First submitted 2021-03-10; First posted 2021-03-15 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2022-08

CONDITIONS: Developmental Disability
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent coaching (Experimental): The parent-coaching intervention consists of up to 8 weekly/fortnightly sessions, and each session will last up to one hour.
  Interventions: Behavioral: Occupational Performance coaching
- Parent consultation (Active Comparator): The parent consultations are given for up to 8 weekly/fortnightly sessions, and each session may last up to one hour.
  Interventions: Behavioral: Parent consultation

INTERVENTIONS:
Behavioral: Occupational Performance coaching — The OPC intervention comprises three components: (1) connect - building parents' trust in the coach by using verbal and nonverbal strategies; (2) structure - building parents' competence by adopting a problem-solving framework of setting goals, exploring options, planning action, carrying out plans, checking performance, and generalizing; and (3) share - building parents' autonomy by reciprocally exchanging information between the coach and parents with an emphasis on eliciting parents existing knowledge. During the exploration of the options for a particular goal, collaborative performance analysis is used. The coach follows the four steps to (a) identify parents' perception of what currently happens, (b) identify what they would like to happen, (c) explore barriers and bridges to the desired performance, and (d) identify their needs for taking actions to achieve goals. Parents are guided to find strategies to facilitate their child's performance to support goal achievement.
  Other Names: OPC
  Arms: Parent coaching
Behavioral: Parent consultation — The parent consultation consists of the use of the toolbox to provide parents with available environmental resources and strategies to enhance community participation of their child with developmental disability, followed by the understanding of current situation and the identification of problems encountered by parents. Direct informing approach will be used to instruct parents about the availability of environmental resources close to their living areas and what they can plan to do by using possible supportive strategies. In addition, information about child disability and/or developmental milestone may be provided if needed.
  Arms: Parent consultation

SUMMARY:
Participation in community activities allows children to meet friends, learns new skills, fosters independence, and paves the foundation for lifelong health. High rates of community participation restriction have been reported in children with developmental disabilities who are aged six years or below, a critical developmental period.

Occupational Performance Coaching (OPC), grounded in self-determination theory, is aimed to facilitate children's participation in life situations through coaching parents. Studies have shown that OPC is effective to promote children's activity participation. However, there have been limited randomized controlled trials demonstrating the efficacy of OPC, especially with the specific focus on children's community participation.

The investigators propose to evaluate the feasibility and acceptability of conducting a pilot randomized controlled trial of OPC for parents of preschool children with developmental disabilities in Hong Kong, and to test its initial efficacy on promoting children's community participation.

DETAILED DESCRIPTION:
Parent coaching emerges as a preferred approach for enhancing performance and participation of children with developmental disabilities (DD), but limited clinical trials examine its effects on community participation. Thus, this study aims to evaluate whether parent coaching, specifically using Occupational Performance Coaching (OPC), enhances community participation among young children with DD.

Young children with DD will be recruited from preschool-rehabilitation services offered by three non-governmental organisations in Hong Kong. Ethics approval has been obtained from the Human Subjects Ethics Sub-committee at The Hong Kong Polytechnic University.

A two-arm parallel, double-blind design will be adopted for the study. Fifty parents of young children with DD will be randomly assigned to the intervention group (i.e., OPC) or the active control group (i.e., parents' consultation). Four assessment points will be scheduled throughout the study: 5-6 weeks before intervention (Time 0), 1-2 weeks before intervention (Time 1), 1-2 weeks after intervention (Time 2), and 8-9 weeks after the intervention (Time 3). Randomisation allocation will be completed at Time 1. Participants and independent outcome assessors will not be informed about the groupings.

Each parent will receive a maximum of eight coaching sessions or consultations. The primary outcome will be children's community participation as assessed through parent-report measures at baseline, pre-intervention, post-intervention, and an 8-week follow-up. Children in both groups will continue to receive their usual care, which may include services such as occupational therapy, physiotherapy, and speech therapy on a weekly/monthly basis, depending on their individual needs.

Independent t-test and chi-square statistics will be used to test for between-group baseline differences. To evaluate the effect of OPC on each outcome measure, repeated-measures analysis of covariance (ANCOVA) by controlling for baseline values per outcome will be used. Post-hoc analyses will be performed when the main effects were significant. Statistical significance is set at p < 0.05. Estimates of effect sizes with 95% confidence intervals will be calculated for each outcome measure.

ELIGIBILITY:
Inclusion Criteria:

* the child has a clinical diagnosis of developmental disability (including but not limited to intellectual disability, developmental delay, or autism spectrum disorder) given by pediatricians/psychiatrist
* the parents are the child's main caregiver who have a long-term parenting role with at least 50% of caregiving responsibilities
* the parents are able to converse in Chinese
* the parents desire to improve their child's participation in community activities

Exclusion Criteria:

* the child has developmental disability combined with physical impairment (e.g., amputation, cerebral palsy, spina bifida)
* the child has developmental disability combined with sensory impairment (e.g., blindness, deafness)

Ages: 24 Months to 83 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Wen Chien, Principal Investigator — The Hong Kong Polytechnic University
Locations (3):
- Hong Kong (3):
  - Hong Kong Christian Service, Kowloon
  - Heep Hong Society, Kwun Tong
  - SAHK, North Point

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chien CW, Lai YYC, Lin CY, Graham F. Occupational Performance Coaching With Parents to Promote Community Participation of Young Children With Developmental Disabilities: Protocol for a Feasibility and Pilot Randomized Control Trial. Front Pediatr. 2021 Nov 5;9:720885. doi: 10.3389/fped.2021.720885. eCollection 2021. PMID 34805034

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Young children with DD were recruited from preschool-rehabilitation services offered by three non-governmental organisations. Two-hundred-and-thirty-six invitations were distributed to interested parents, 61 who were interested for research participation and were then screened, and 50 whose children met the eligible criteria participated in the RCT.
Pre-assignment Details: Out of the 61 parents who underwent eligibility screening, five did not meet inclusion criteria and six declined to participate. The 50 parents and their children (i,e., 50 dyads) were finally enrolled in this study.
Period: Overall Study
Arm/Group | Parent Coaching | Parent Consultation
Started | 25 (Children = 25, Parents = 25) | 25 (Children = 25, Parents = 25)
Completed | 24 (Children = 24, Parents = 24) | 24 (Children = 24, Parents = 24)
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Parent Coaching: Parents received OPC
- Parent Consultation: Parents received consultation
- Total: Total of all reporting groups
Arm/Group | Parent Coaching | Parent Consultation | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25 | 25 | 50
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Children Population: The analysis was conducted separately for children and parents.
  years
    Children: number analyzed (Participants) | 25 | 25 | 50
    Children | 4.85 (1.00) | 4.82 (0.96) | 4.83 (1.0)
    Parents: number analyzed (Participants) | 25 | 25 | 50
    Parents | 35.92 (5.99) | 39.44 (3.72) | 37.68 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants] — Children Population: The analysis was conducted separately for children and parents.
  Participants
    Children: number analyzed (Participants) | 25 | 25 | 50
    Children: Female | 10 | 9 | 19
    Children: Male | 15 | 16 | 31
    Parents: number analyzed (Participants) | 25 | 25 | 50
    Parents: Female | 24 | 23 | 47
    Parents: Male | 1 | 2 | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Hong Kong | 50 | 50 | 100
Community-related goal performance for children [Mean (Standard Deviation); unit: units on a scale] — The Canadian Occupational Performance Measure (COPM) measures parents' perceptions of children's participation in specific community activities. Parents are prompted to rate their child's performance on a 10-point Likert scale (1 = not good at all and 10 = optimal performance). Average scores (1-10) can be generated, and high scores indicate greater children's participation performance. Population: This measure was collected for child performance related to the community-related goal. There were no results from parents' performance.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 3.67 (1.66) | 3.72 (1.39) | 3.69 (1.52)
Community-related goal satisfaction for parents [Mean (Standard Deviation); unit: units on a scale] — The Canadian Occupational Performance Measure (COPM) measures parents' perceptions of children's participation in specific community activities. Parents are prompted to rate their satisfaction with the current status on a 10-point Likert scale (1 = not satisfied at all and 10 = optimal satisfaction). Average scores (1-10) can be generated, and high scores indicate greater parents' satisfaction. Population: This measure was collected for parents' satisfaction on the community-related goal for their children. There were no results from children's satisfaction.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 3.90 (1.62) | 3.57 (1.45) | 3.73 (1.53)
Community participation frequency for children [Mean (Standard Deviation); unit: units on a scale] — The Young Children's Participation and Environment Measure (YC-PEM) capture children's overall community participation patterns. It has a community section that includes 11 participation items and parents are asked to rate how often their child has participated in the past four months using an 8-point Likert scale (0 = never and 7 = once or more each day). Average scores (0-7) can be generated, and high scores indicate greater children's participation frequency. Population: This measure collected only the frequency of children's participation in community activities. No data were collected for parents.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 3.02 (0.79) | 2.74 (0.90) | 2.88 (0.85)
Community participation involvement for children [Mean (Standard Deviation); unit: units on a scale] — The Young Children's Participation and Environment Measure (YC-PEM) capture children's overall community participation patterns. It has a community section that includes 11 participation items and parents are asked to rate how involved the child is during participation using a 5-point Likert scale (1 = not very involved and 5 = very involved). Average scores (1-5) can be generated, and high scores indicate greater children's participation involvement. Population: This measure collected only children's participation involvement in community activities. No data were collected for parents.
  units on a scale
    number analyzed (Participants) | 25 | 25 | 50
    (all) | 3.85 (0.77) | 3.77 (0.72) | 3.81 (0.74)

OUTCOME MEASURES:

1. Primary Outcome: Change in Participation-related Goal Performance and Satisfaction
Description: Performance and satisfaction scores (1-10) of the Canadian Occupational Performance Measure (COPM). Higher scores mean a better outcome.
Time Frame: T0=5-6 weeks before intervention; T1=1-2 weeks before intervention; T2=1-2 weeks after intervention; T3=8-9 weeks after the intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale
  Performance at T0 | 3.67 (1.66) | 3.72 (1.39)
  Performance at T1 | 4.92 (1.73) | 4.69 (1.70)
  Performance at T2 | 7.29 (1.49) | 6.85 (1.63)
  Performance at T3 | 7.16 (1.30) | 6.84 (1.68)
  Satisfaction at T0 | 3.90 (1.62) | 3.57 (1.45)
  Satisfaction at T1 | 4.85 (1.87) | 4.68 (1.84)
  Satisfaction at T2 | 7.58 (1.39) | 7.08 (1.71)
  Satisfaction at T3 | 7.32 (1.33) | 6.84 (1.82)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, Repeated-measures ANCOVA

2. Primary Outcome: Change in Children's Community Participation Frequency and Involvement
Description: Frequency scores (0-7) and involvement scores (1-5) of the community section of the Young Children's Participation and Environment Measure (YC-PEM). Higher scores mean a better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale
  Community frequency at T0 | 3.02 (0.79) | 2.74 (0.90)
  Community frequency at T1 | 3.14 (0.83) | 2.79 (1.12)
  Community frequency at T2 | 3.35 (1.00) | 2.81 (1.06)
  Community frequency at T3 | 3.42 (1.18) | 2.91 (0.95)
  Community involvement at T0 | 3.85 (0.77) | 3.77 (0.72)
  Community involvement at T1 | 3.77 (0.69) | 3.82 (0.83)
  Community involvement at T2 | 4.12 (0.53) | 4.13 (0.69)
  Community involvement at T3 | 4.08 (0.64) | 4.15 (0.70)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, Repeated-Measures ANCOVA

3. Secondary Outcome: Change in Parenting Efficacy and Satisfaction
Description: Efficacy scores (7-42) and satisfaction scores (9-56) of the Parenting Sense of Competence Scale (PSOC). Higher scores mean a better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale
  Parenting efficacy at T0 | 27.52 (5.81) | 27.92 (3.82)
  Parenting efficacy at T1 | 27.76 (6.06) | 27.52 (4.54)
  Parenting efficacy at T2 | 29.44 (5.47) | 30.48 (3.94)
  Parenting efficacy at T3 | 28.76 (5.78) | 29.28 (4.87)
  Parenting satisfaction at T0 | 31.60 (7.37) | 31.56 (8.20)
  Parenting satisfaction at T1 | 30.72 (8.38) | 32.40 (8.69)
  Parenting satisfaction at T2 | 33.80 (6.67) | 33.16 (7.80)
  Parenting satisfaction at T3 | 31.76 (8.08) | 33.32 (8.07)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, Repeated-Measures ANCOVA

4. Secondary Outcome: Change in Parents' Negative Emotional States
Description: The scores (0-42 for each subscale) of the Depression, Anxiety and Stress Scale-21 (DASS-21). Higher scores mean a worse outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale
  Depression at T0 | 7.04 (6.78) | 10.00 (10.39)
  Depression at T1 | 7.28 (8.03) | 10.56 (11.51)
  Depression at T2 | 6.32 (7.11) | 9.04 (11.28)
  Depression at T3 | 6.56 (7.38) | 8.40 (10.08)
  Anxiety at Time 0 | 6.80 (5.83) | 10.88 (10.53)
  Anxiety at T1 | 6.96 (7.89) | 10.64 (10.24)
  Anxiety at T2 | 6.08 (7.10) | 10.00 (11.81)
  Anxiety at T3 | 6.48 (7.19) | 8.88 (10.00)
  Stress at T0 | 15.12 (10.67) | 14.64 (10.65)
  Stress at T1 | 15.04 (12.55) | 16.44 (10.18)
  Stress at T2 | 13.92 (11.96) | 16.00 (10.59)
  Stress at T3 | 14.40 (11.78) | 13.76 (9.83)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, Repeated-Measures ANCOVA

5. Secondary Outcome: Change in Children's Psychosocial Health
Description: Psychosocial health score (0-100) of the KINDL questionnaire. Higher scores mean a better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale
  Psychological health at T0 | 67.50 (10.52) | 66.50 (11.84)
  Psychological health at T1 | 66.68 (12.69) | 65.00 (7.90)
  Psychological health at T2 | 70.00 (12.52) | 67.81 (10.33)
  Psychological health at T3 | 67.50 (10.52) | 65.50 (11.84)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, Repeated-Measures ANCOVA

6. Other Pre Specified Outcome: Stability in Children's Daily Activity and Social/Cognitive Function
Description: Scaled scores (0-100) of the daily activity and social/cognitive domains of the Pediatric Evaluation of Disability Inventory computer-adaptive tests (PEDI-CAT). Higher scores mean a better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale
  Daily activity at T0 | 57.12 (4.77) | 56.40 (2.98)
  Daily activity at T1 | 57.52 (4.81) | 56.48 (3.53)
  Daily activity at T2 | 59.16 (3.92) | 58.04 (3.44)
  Daily activity at T3 | 59.08 (4.27) | 58.12 (3.50)
  Social/cognitive function at T0 | 64.96 (3.06) | 63.56 (3.45)
  Social/cognitive function at T1 | 64.84 (3.54) | 63.92 (2.87)
  Social/cognitive function at T2 | 66.40 (3.09) | 65.80 (3.36)
  Social/cognitive function at T3 | 66.56 (3.72) | 66.12 (3.00)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, Repeated-Measures ANCOVA

7. Other Pre Specified Outcome: Stability in Perceived Impact of Environmental Support on Children's Community Participation
Description: Perceived environmental support scores (0-100) of the community section of the Young Children's Participation and Environment Measure. Higher scores mean a better outcome.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale
  Environmental support at T0 | 84.07 (9.62) | 78.11 (11.35)
  Environmental support at T1 | 83.84 (11.65) | 80.70 (10.40)
  Environmental support at T2 | 85.07 (11.49) | 83.29 (11.35)
  Environmental support at T3 | 84.86 (8.72) | 80.31 (11.73)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, Repeated-Measures ANCOVA

8. Other Pre Specified Outcome: Level of Therapeutic Alliance During Coaching Session
Description: Total scores (0-40) of the Session Rating Scale (SRS). Higher average scores mean a better outcome.
Time Frame: Immediate after each of the coaching sessions during the intervention period
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale | 35.28 (4.63) | 36.53 (4.09)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, t-test, 2 sided

9. Other Pre Specified Outcome: Level of Perceptions of Health Care Practitioners' Autonomy Support
Description: Total scores (1-7) of the Health Care Climate Questionnaire (HCCQ). Higher scores mean a better outcome.
Time Frame: T1=1-2 weeks before intervention; T2=1-2 weeks after intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
score on a scale
  T1 | 5.58 (0.94) | 5.62 (0.93)
  T2 | 5.72 (0.90) | 6.12 (0.85)
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, t-test, 2 sided

10. Other Pre Specified Outcome: Level of Parents' Global Impression on the Improvement of Their Child's Community Participation
Description: The item score (1-7) of the Patient Global Impression of Change. Higher scores mean a worse outcome.
Time Frame: T2=1-2 weeks after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
Participants
  Very much improved | 3 | 5
  Much improved | 8 | 6
  A little improved | 11 | 12
  No change | 3 | 1
  A little deterioration | 0 | 1
  Much deterioration | 0 | 0
  Very much deterioration | 0 | 0
Statistical Analysis 1: Comparison: Parent Coaching vs Parent Consultation; Test type: Superiority; p = 0.05, Chi-squared

11. Other Pre Specified Outcome: Number of Participants Recruited
Description: The percentage of eligible families agreeing to participate in the study
Time Frame: T0=5-6 weeks before intervention
Measure: Count of Participants; unit: Participants
Groups:
- Total Group: Two groups were merged into one total group for calculation
Arm/Group | Total Group
Number analyzed (Participants) | 236
Participants | 50

12. Other Pre Specified Outcome: Retention Rate of Participants Who Complete the Trial
Description: The percentage of participants who complete the trial (i.e., all assessments)
Time Frame: T3=8-9 weeks after the intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
Participants | 24 | 25

13. Other Pre Specified Outcome: Adherence Rate of Participants Who Attend the Coaching Sessions
Description: The percentage of coaching sessions attended by parents who are randomized to the intervention group
Time Frame: T2=1-2 weeks after intervention
Measure: Count of Units; unit: Number of sessions
Units Other Than Participants: Number of sessions
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
Number analyzed (Number of sessions) | 200 | 200
Number of sessions | 171 | 192

14. Other Pre Specified Outcome: Blinding Success
Description: The percentage of parents who guess treatment allocation correctly after the study
Time Frame: T2=1-2 weeks after intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Coaching | Parent Consultation
Number analyzed (Participants) | 25 | 25
Participants | 8 | 16

15. Other Pre Specified Outcome: Fidelity of Coaches Who Conduct the Occupational Performance Coaching
Description: Percentage score of the Occupational Performance Coaching Fidelity Measure. This measure consists of 18 items across five domains: relationship, goal, reflection, analysis and action, client response, and distinguishing. Each item is rated on a three-point Likert scale (1 = low and 3 = high). The percentage score can be calculated by dividing the total score by the possible maximum score. Higher percentage scores indicate higher fidelity, and the cut-off of sufficient fidelity of coaching per session is set at 80%.
Time Frame: T2=1-2 weeks after intervention
Measure: Count of Participants; unit: Participants
Groups:
- Parent Coaching: Coaching fidelity was calculated only for the parent coaching group
Arm/Group | Parent Coaching
Number analyzed (Participants) | 8
Participants | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected usually during the intervention period; that is, 4 months.
Description: Both parents and children were monitored/assessed in this study.
Groups:
- Parent Coaching - Parent Participants; Parent Coaching - Children Participants: The parent-coaching intervention consists of up to 8 weekly/fortnightly sessions, and each session will last up to one hour.
  Occupational Performance coaching: The OPC intervention comprises three components: (1) connect - building parents' trust in the coach by using verbal and nonverbal strategies; (2) structure - building parents' competence by adopting a problem-solving framework of setting goals, exploring options, planning action, carrying out plans, checking performance, and generalizing; and (3) share - building parents' autonomy by reciprocally exchanging information between the coach and parents with an emphasis on eliciting parents existing knowledge. During the exploration of the options for a particular goal, collaborative performance analysis is used. The coach follows the four steps to (a) identify parents' perception of what currently happens, (b) identify what they would like to happen, (c) explore barriers and bridges to the desired performance, and (d) identify their needs for taking actions to achieve goals. Parents are guided to find strategies to facilitate their child's performance to support goal achievement.
- Parent Consultation - Parent Participants; Parent Consultation - Children Participants: The parent consultations are given for up to 8 weekly/fortnightly sessions, and each session may last up to one hour.
  Parent consultation: The parent consultation consists of the use of the toolbox to provide parents with available environmental resources and strategies to enhance community participation of their child with developmental disability, followed by the understanding of current situation and the identification of problems encountered by parents. Direct informing approach will be used to instruct parents about the availability of environmental resources close to their living areas and what they can plan to do by using possible supportive strategies. In addition, information about child disability and/or developmental milestone may be provided if needed.
Arm/Group | Parent Coaching - Parent Participants | Parent Coaching - Children Participants | Parent Consultation - Parent Participants | Parent Consultation - Children Participants
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25 | 0/25

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic posed significant challenges, impacting the intervention delivery and outcomes across all measures. The study's sample size was small and also excluded children with physical impairments. Two therapists fell short of achieving the stipulated 80% coaching fidelity in their initial cases and were not assigned further cases. Convenience sampling was used for participant recruitment, and families who chose to participate might have higher motivation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-22): https://cdn.clinicaltrials.gov/large-docs/09/NCT04796909/Prot_SAP_000.pdf